CLINICAL TRIAL: NCT07244757
Title: Comparison of Two Dosing Regimens of Intravenous Ketorolac for Post-Cesarean Pain Control: A Randomized Controlled Trial
Brief Title: Comparison of Two Dosing Regimens of Intravenous Ketorolac for Post-Cesarean Pain Control
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MS-390-2025
Record Dates: First submitted 2025-11-16; First posted 2025-11-24 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Analgesia; Cesarean Delivery; Ketorolac
MeSH Terms: interventions — Ketorolac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ketorolac 30 (Active Comparator): patients will receive intravenous ketorolac at 30 mg/8 h postoperatively
  Interventions: Drug: Ketorolac 30 mg
- ketorolac 15 mg (Active Comparator): patients will receive intravenous ketorolac at 15 mg/8 h postoperatively
  Interventions: Drug: Ketorolac 15mg

INTERVENTIONS:
Drug: Ketorolac 30 mg — administered intravenously as 30 mg diluted in 10 mL of normal saline and injected over more than 15 seconds
  Arms: ketorolac 30
Drug: Ketorolac 15mg — administered intravenously as either 15 mg diluted in 10 mL of normal saline and injected over more than 15 seconds.
  Arms: ketorolac 15 mg

SUMMARY:
we aim to compare the analgesic efficacy of two intravenous ketorolac dosing regimens as part of a multimodal analgesic protocol that includes local wound infiltration for postoperative pain management after elective cesarean delivery.

DETAILED DESCRIPTION:
Spinal anesthesia will be achieved by injecting 10 mg hyperbaric bupivacaine 0.5% plus 25 mcg fentanyl Prophylactic vasopressor will be administered in all patients, Following delivery, all patients will receive a single dose of dexamethasone (8 mg) along with the first dose of intravenous ketorolac. Subsequent ketorolac doses will be administered every 8 hours.

After closing the fascia, the subcutaneous layer will be infiltrated with 30 mL of 0.25% bupivacaine.

Postoperatively, if the Numeric rating scale is > 3, intravenous nalbuphine 0.1 mg/kg titrated to response, with maximum single dose of 20 mg and maximum daily dose of 160 mg.

ELIGIBILITY:
Inclusion Criteria:

* full-term, singleton, pregnant women,
* aged 18-35 years,
* scheduled for elective cesarean delivery under spinal anesthesia

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) physical class III or more
* multiple gestation. Patients with a history of allergy to any of the study drugs,
* renal impairment,
* gastrointestinal bleeding or ulceration
* inflammatory bowel disease,
* chronic pain or regular opioid use.
* Inability to comprehend the numeric pain scale (NRS) or the ObsQoR-11 score
* requirement for conversion to general anesthesia after spinal anesthesia

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
numeric rating scale at rest | 6 hours postoperatively
  the patient rates their pain on a scale of 0 to 10, with 0 being "no pain" and 10 being the "worst pain imaginable"

SECONDARY OUTCOMES:
numeric rating scale at rest | at 30 minutes, 12-, 18-, and 24 hours postoperatively
  person rates their pain on a scale of 0 to 10, with 0 being "no pain" and 10 being the "worst pain imaginable"
numeric rating scale during movement | at 30 minutes, 6-, 12-, 18-, and 24 hours postoperatively
  person rates their pain on a scale of 0 to 10, with 0 being "no pain" and 10 being the "worst pain imaginable" during change position from supine to sitting or ambulation
total nalbuphine consumption | from 0.5 hour postoperatively to 24 hour postoperatively
  mg
time to first analgesic requirement | time from immediately postoperatively to time of first analgesic requirement during the first 24 hours
  hours
ObsQoR-11 score | 24 hour postoperatively
  The ObsQoR-11 is an 11-item questionnaire to assess a patient's recovery after a C-section, with a total score ranging from 0 to 100, where 100 is the best possible recovery
patient's satisfaction | 24 hour postoperatively
  At the end of the study the patient will be asked to rate her satisfaction with pain control using the NRS 10= strongly unsatisfied, 0= strongly satisfied

CONTACTS AND LOCATIONS:
Overall Officials: ahmed hasanin, Principal Investigator — Cairo University Kasr Alainy Faculty of Medicine
Locations (1):
- Kasr Alainy Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
data used for analysis will be available from the PI upon reasonable requist
Supporting Information: Study Protocol, SAP